CLINICAL TRIAL: NCT06201975
Title: Efficacy of Locally Delivered Thyme Honey as a Novel Adjunct to Non-surgical Periodontal Therapy: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Thyme Honey as a Novel Adjunct to Non-surgical Periodontal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Dalia Ghalwash, Professor anf Head of department, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-062
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Diseases
Keywords: Periodontitis; Thyme honey; anti-inflammatory
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: The experimental group will receive scaling and root debridement and locally delivered 0.5 ml non-diluted Thyme honey on sites with PPD ≥ 5 mm. Thyme honey will be delivered to the sites until overflows using a syringe with plastic catheter of cannula 20 g (B Braun) attached to it. Patients will be reviewed at 6 weeks to re-evaluate the clinical periodontal parameters.
  The control group will receive scaling and root debridement with normal saline irrigation on sites with PPD ≥ 5 mm.
Who Masked: Outcomes Assessor
Masking Description: The clinical outcome assessor (A.A) will not be aware of which treatment will be being administered, thus yielding a single-blind controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyme honey (Experimental): The experimental group will receive scaling and root debridement and locally delivered 0.5 ml non-diluted Thyme honey on sites with PPD ≥ 5 mm. Thyme honey will be delivered to the sites until overflows using a syringe with plastic catheter of cannula 20 g (B Braun) attached to it. Patients will be reviewed at 6 weeks to re-evaluate the clinical periodontal parameters (Ibrahim et al., 2021).
  Interventions: Other: Thyme honey
- Saline (Placebo Comparator): The control group will receive scaling and root debridement with normal saline irrigation on sites with PPD ≥ 5 mm.
  Interventions: Other: Thyme honey

INTERVENTIONS:
Other: Thyme honey — Thyme honey will be delivered to the sites until overflows using a syringe with plastic catheter of cannula 20 g (B Braun) attached to it. Patients will be reviewed at 6 weeks to re-evaluate the clinical periodontal parameters

SUMMARY:
Periodontal diseases are disease processes involving the periodontium, a term used to describe the supportive apparatus surrounding the tooth, which includes the gingival tissue, alveolar bone, cementum, and periodontal ligament. Thyme honey, as a conventional therapy, might be a novel antioxidant to abate many of the diseases directly or indirectly associated with oxidative stress. To the best of the researchers' knowledge, there are no published studies on the management of periodontitis in using locally delivered Thyme honey.

DETAILED DESCRIPTION:
In 2017, the American Academy of Periodontology, in collaboration with the European Federation of Periodontology, devised a new classification of periodontal and peri-implant diseases. In this new classification, periodontitis can be subdivided into three categories, Necrotizing periodontal diseases, Periodontitis, Periodontitis as a manifestation of systemic diseases.

Non-surgical treatment is valuable in mild to moderate periodontitis whereas surgical treatment is useful in progressive cases. Confined drug delivery systems-mouth rinses, irrigating solutions and sustained release devices are used for distribution of antimicrobial agents.

It has been observed that artificial antimicrobial agents and antibiotics are identified to cause antimicrobial resistance. It has also been observed that appearance of formerly rare infections is on the rise perhaps due to the incorrect or prevalent overuse of antimicrobials. Natural phytochemicals have demonstrated to be worthy substitutes to synthetic agents.

It is interesting fact to note that two of the most populated countries in the world China and India, have used herbal medicine for the managing of oral infections, comprising periodontal disease as well for more than a duration of 2000 years.

It has been found that in adults with chronic periodontitis, scaling and root planning along with use of an adjunctive antimicrobial mediator increases patient outcomes over a period of time compared to scaling alone. Modern chemotherapeutic agents display significant efficacy in improving periodontal health but owing to undesirable side effects such as tooth discoloration, taste alteration, and price of these substances, the usage of herbal products has increased lately and could be especially of high benefit to lower socioeconomic populations around the world.

Herbal medicines and preparations comprise of plant constituents professed to have therapeutic benefits. Herbal products are favored over conventional drugs owing to extensive natural activity, advanced safety margin, and inferior costs. Additionally, the modern drugs are known to cause several side effects. Continuous intake of modern drugs has sometimes caused in antibiotic resistance thereby herbal medicines are being used gradually as dietary add-ons to combat or avert common ailments affecting human body and oral cavity.

Honey as a natural product has clinched the attention of researchers as a complementary and alternative medicine. Honey as a folk medicine is referred in the utmost ancient written archives.

Demarcation of its uses in current professional medicine as a potential therapy is entirely underutilized. However, there is an affinity for some researchers to fire out a coherent proposition that usage of honey as a natural product supplement is well intentioned for reflection as a therapy or adjuvant antioxidant therapy in current medicine. The composition of honey varies from floral source to origin.

Thyme honey has been studied against various ailments in animal and human models. Published research denotes it as a novel antioxidant agent. It exhibits a broad spectrum therapeutic properties such as anti-inflammatory, antibacterial, antimutagenic, expedite wound healings, antidiabetic, antiviral, antifungal, and antitumor effects.

Additionally, the anti-inflammatory properties of Greek thymus vulgaris extract was examined in recent research which reported its ability to reduce the LPS-induced elevation in cyclooxygenase (COX)-2, nuclear factor-kappa B (NF-кB), TNF-α, and produced a more potent attenuating effect than dexamethasone for most of the studied inflammatory mediators.

Moreover, thymol was reported to possess an inhibitory effect on TNF-α, IL-6, IFN-γ, IL-1β and IL-17, C-reactive protein and myeloperoxidase. Furthermore, unfractionated essential oil from T. vulgaris was found to reduce neutrophil infiltration during inflammatory response.Thyme honey, as a conventional therapy, might be a novel antioxidant to abate many of the diseases directly or indirectly associated with oxidative stress. To the best of the researchers' knowledge, there are no published studies on the management of periodontitis in using locally delivered Thyme honey.

ELIGIBILITY:
Inclusion Criteria:

* - Both genders, aged above 18 years.
* All patients must have a periodontal disease.
* Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol.
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment loss (CAL) | 6 weeks
  With a periodontal probe, PD and CAL will be measured on six locations of the teeth (mesio-buccal/facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal).

SECONDARY OUTCOMES:
Bleeding on probing | 6 weeks
  The proportion of bleeding sites 10 second after being stimulated by a standardized manual probe with a controlled force to the bottom of the sulcus/pocket at six locations (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual) on all present teeth will be assessed dichotomously as a BOP score on all present teeth